CLINICAL TRIAL: NCT05771324
Title: The Effect of Baby-Led Weaning and Traditional Complementary Feeding Education on Infant Development Randomized Controlled Trial
Brief Title: The Effect of Baby-Led Weaning and Traditional Complementary Feeding Education on Infant Development
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Nurten ARSLAN, lecturer, Zonguldak Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: nurten.arslan; 2020-19093093-02 (Other Grant/Funding Number: Zonguldak Bulent Ecevit University)
Record Dates: First submitted 2023-02-05; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Growth; Infant Development; Complementary Feeding; Nutrition, Healthy; Anemia, Iron Deficiency; Obesity, Infant
Keywords: Growth; Infant Development; Complementary Feeding; Nutrition, Healthy; Anemia, Iron Deficiency; Obesity, Infant; solid food
MeSH Terms: conditions — Anemia, Iron-Deficiency; Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: The sample size of the study consisted of 62 people according to the power analysis. Block and stratified randomization methods were used in the selection of the experimental groups. When the literature is examined, there are studies showing the effect of mothers' education level and previous complementary food experiences on the transition to solid food. Accordingly, stratification was made according to the education level of the mothers and the number of children. Thus, two people were assigned homogeneously in each block according to the education level of the mothers and the number of children. Randomization was done by the Outcome Evaluator independently of the investigators. The research was carried out according to the Consort 2010 Flow Chart and the study was concluded with 56 people.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participants who were assigned to the researcher groups that evaluated the hematological test results of the babies and followed the growth were kept confidential from the interventions.
  The person evaluating the outcomes was kept confidential from the participant and the interventions.
  Participants did not know about the other intervention group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baby-Led Weaning (BLW) (Experimental): The group named for infants who received complementary feeding education with the BLW method and who were fed with the BLW method.
  Interventions: Other: Baby-Led Weaning (BLW)
- Traditional Complementary Feeding (TCF) (Experimental): The group named for infants who received complementary nutrition education with the TCF method and who were fed with the TCF method.
  Interventions: Other: Traditional Complementary Feeding (TCF)

INTERVENTIONS:
Other: Baby-Led Weaning (BLW) — BLW trainings given to mothers for 6-12 month old babies
  Other Names: BLW
  Arms: Baby-Led Weaning (BLW)
Other: Traditional Complementary Feeding (TCF) — TCF trainings given to mothers for 6-12 month old babies
  Other Names: TCF
  Arms: Traditional Complementary Feeding (TCF)

SUMMARY:
The goal of this [type of study: clinical trial] is to compare compare the nutrition, development, obesity risk and anemia risk of the infant with the BLW method and TCF method given to the mothers of infants who have switched to complementary feeding. The main question[s] it aims to answer are:

* Does the training on the GTB and BLW method given in accordance with the developmental age of the baby in months have an effect on the feeding and development of the babies in both groups?
* Does the training on the GTB and BLW method given in accordance with the developmental age of the baby in months have an effect on the obesity risk and anemia risk of babies in both groups?

Participants will participate in each session of the complementary nutrition trainings given in accordance with their age on a monthly basis and will provide a diet suitable for the trainings.

Researchers will compare the nutritional parameters, developmental levels, and height and weight gains of infants fed with the BLW and TCF method to see the effect of complementary feeding education on the nutrition and development of infants and whether there is anemia and obesity risk.

DETAILED DESCRIPTION:
Regarding the basic questions that the study aims to answer;

Micronutrient intake, hemoglobin, ferritin and vitamin B12 levels were evaluated to examine the effects of the trainings on infant nutrition.

Physical, cognitive, psychosocial, language, motor and game development levels of infants were evaluated in order to examine the effects of training on infant development.

Weight gain, WLZ, LAZ and WAZ scores of infants were evaluated to examine the effects of the education given on obesity risk.

Hemoglobin, hematocrit and ferritin levels were evaluated to examine the effects of the training given on the risk of anemia.

ELIGIBILITY:
Inclusion Criteria:

for mothers;

* The fact that the mothers came to the center where the research will be conducted for routine baby follow-up and vaccination follow-up.
* Mothers' willingness to participate in the research
* Absence of any communication problems
* The mothers must be at least 19 years old.
* Mothers have no physical or mental disability

for babies;

. Babies must be at least 4 months and maximum 6 months old when they are included in the study.

* Complementary feeding not yet started
* Babies being fed only with breast milk
* Babies not born before 38 weeks of gestation
* Absence of a congenital anomaly
* Absence of any digestive and neurological system diseases that may affect nutrition

Exclusion Criteria:

* Infants and mothers who did not meet the inclusion criteria were not included in the study.

Ages: 4 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2021-04-18 (Actual); Study Completion 2022-04-18 (Actual)

PRIMARY OUTCOMES:
Effect on infant growth | Examining the change at 12 months
  BMI of babies were used as growth criteria. In addition, Z-score values for BMI were examined according to WHO standards.
Effect on infant developmenter parameter | Examining the change at 12 months
  In the evaluation of infant development, motor developmental evaluation criteria used as standard in the national infant follow-ups of the T.C. Ministry of Health were used.
Effect on infant anemia and iron deficiency | Examining the change at 12 months.
  Iron levels in infants were examined.
Effect on infant obesity risk | Examining the change at 12 months.
  The 12-month BMI distributions of the groups were analyzed.

SECONDARY OUTCOMES:
Early transition to solid food | Examining the change at 12 months.
  Solid food intake time in infants in both groups was evaluated as months
Early transition to self feeding | Examining the change at 12 months
  Self feeding time in infants in both groups was evaluated as months
Early transition to family meals | Examining the change at 12 months.
  Family meals time in infants in both groups was evaluated as months

CONTACTS AND LOCATIONS:
Overall Officials: NURTEN ARSLAN, Principal Investigator — Zonguldak Bulent Ecevit University
Locations (1):
- ZonguldakBEU, Zonguldak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The researcher who made the evaluation did not have information about the experimental groups and which group the individuals were assigned to.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data can be shared immediately after summary data is published.
Access Criteria: The data were shared with the statistician for analysis.

REFERENCES:
- [Background] Cameron SL, Taylor RW, Heath AL. Development and pilot testing of Baby-Led Introduction to SolidS--a version of Baby-Led Weaning modified to address concerns about iron deficiency, growth faltering and choking. BMC Pediatr. 2015 Aug 26;15:99. doi: 10.1186/s12887-015-0422-8. PMID 26306667
- [Background] Cameron SL, Taylor RW, Heath AL. Parent-led or baby-led? Associations between complementary feeding practices and health-related behaviours in a survey of New Zealand families. BMJ Open. 2013 Dec 9;3(12):e003946. doi: 10.1136/bmjopen-2013-003946. PMID 24327363
- [Background] Cameron SL, Heath AL, Taylor RW. How feasible is Baby-led Weaning as an approach to infant feeding? A review of the evidence. Nutrients. 2012 Nov 2;4(11):1575-609. doi: 10.3390/nu4111575. PMID 23201835
- [Background] Daniels L, Taylor RW, Williams SM, Gibson RS, Fleming EA, Wheeler BJ, Taylor BJ, Haszard JJ, Heath AM. Impact of a modified version of baby-led weaning on iron intake and status: a randomised controlled trial. BMJ Open. 2018 Jun 27;8(6):e019036. doi: 10.1136/bmjopen-2017-019036. PMID 29950456
- [Background] Daniels L, Heath AL, Williams SM, Cameron SL, Fleming EA, Taylor BJ, Wheeler BJ, Gibson RS, Taylor RW. Baby-Led Introduction to SolidS (BLISS) study: a randomised controlled trial of a baby-led approach to complementary feeding. BMC Pediatr. 2015 Nov 12;15:179. doi: 10.1186/s12887-015-0491-8. PMID 26563757
- [Background] Williams Erickson L, Taylor RW, Haszard JJ, Fleming EA, Daniels L, Morison BJ, Leong C, Fangupo LJ, Wheeler BJ, Taylor BJ, Te Morenga L, McLean RM, Heath AM. Impact of a Modified Version of Baby-Led Weaning on Infant Food and Nutrient Intakes: The BLISS Randomized Controlled Trial. Nutrients. 2018 Jun 7;10(6):740. doi: 10.3390/nu10060740. PMID 29880769
- [Background] Morison BJ, Taylor RW, Haszard JJ, Schramm CJ, Williams Erickson L, Fangupo LJ, Fleming EA, Luciano A, Heath AL. How different are baby-led weaning and conventional complementary feeding? A cross-sectional study of infants aged 6-8 months. BMJ Open. 2016 May 6;6(5):e010665. doi: 10.1136/bmjopen-2015-010665. PMID 27154478
- [Background] Robert RC, Creed-Kanashiro HM, Villasante R, Narro MR, Penny ME. Strengthening health services to deliver nutrition education to promote complementary feeding and healthy growth of infants and young children: formative research for a successful intervention in peri-urban Trujillo, Peru. Matern Child Nutr. 2017 Apr;13(2):e12264. doi: 10.1111/mcn.12264. Epub 2016 Mar 2. PMID 26931182
- [Background] Taylor RW, Williams SM, Fangupo LJ, Wheeler BJ, Taylor BJ, Daniels L, Fleming EA, McArthur J, Morison B, Erickson LW, Davies RS, Bacchus S, Cameron SL, Heath AM. Effect of a Baby-Led Approach to Complementary Feeding on Infant Growth and Overweight: A Randomized Clinical Trial. JAMA Pediatr. 2017 Sep 1;171(9):838-846. doi: 10.1001/jamapediatrics.2017.1284. PMID 28692728
- [Background] Brown A, Lee M. An exploration of experiences of mothers following a baby-led weaning style: developmental readiness for complementary foods. Matern Child Nutr. 2013 Apr;9(2):233-43. doi: 10.1111/j.1740-8709.2011.00360.x. Epub 2011 Nov 28. PMID 22118242
- [Background] Sazawal S, Dhingra P, Dhingra U, Gupta S, Iyengar V, Menon VP, Sarkar A, Black RE. Compliance with home-based fortification strategies for delivery of iron and zinc: its effect on haematological and growth markers among 6-24 months old children in north India. J Health Popul Nutr. 2014 Jun;32(2):217-26. PMID 25076659
- [Background] D'Auria E, Bergamini M, Staiano A, Banderali G, Pendezza E, Penagini F, Zuccotti GV, Peroni DG; Italian Society of Pediatrics. Baby-led weaning: what a systematic review of the literature adds on. Ital J Pediatr. 2018 May 3;44(1):49. doi: 10.1186/s13052-018-0487-8. PMID 29724233
- [Result] ESPGHAN Committee on Nutrition; Agostoni C, Braegger C, Decsi T, Kolacek S, Koletzko B, Michaelsen KF, Mihatsch W, Moreno LA, Puntis J, Shamir R, Szajewska H, Turck D, van Goudoever J. Breast-feeding: A commentary by the ESPGHAN Committee on Nutrition. J Pediatr Gastroenterol Nutr. 2009 Jul;49(1):112-25. doi: 10.1097/MPG.0b013e31819f1e05. PMID 19502997
- [Result] Alvisi P, Brusa S, Alboresi S, Amarri S, Bottau P, Cavagni G, Corradini B, Landi L, Loroni L, Marani M, Osti IM, Povesi-Dascola C, Caffarelli C, Valeriani L, Agostoni C. Recommendations on complementary feeding for healthy, full-term infants. Ital J Pediatr. 2015 Apr 28;41:36. doi: 10.1186/s13052-015-0143-5. PMID 25928205
- [Result] Brown A, Jones SW, Rowan H. Baby-Led Weaning: The Evidence to Date. Curr Nutr Rep. 2017;6(2):148-156. doi: 10.1007/s13668-017-0201-2. Epub 2017 Apr 29. PMID 28596930
- [Result] Brown A. No difference in self-reported frequency of choking between infants introduced to solid foods using a baby-led weaning or traditional spoon-feeding approach. J Hum Nutr Diet. 2018 Aug;31(4):496-504. doi: 10.1111/jhn.12528. Epub 2017 Dec 5. PMID 29205569
- [Derived] Arslan N, Kurtuncu M, Turhan PM. The effect of baby-led weaning and traditional complementary feeding trainings on baby development. J Pediatr Nurs. 2023 Nov-Dec;73:196-203. doi: 10.1016/j.pedn.2023.09.006. Epub 2023 Sep 13. PMID 37714048